CLINICAL TRIAL: NCT04161716
Title: Study Evaluating the Ability of a NIRS Module to Detect a Urodynamic Variation in Humans
Brief Title: Study Evaluating the Ability of a NIRS Module to Detect a Urodynamic Variation in Humans (DETTECH)
Acronym: DETTECH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BioSerenity (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 2019-A02770-57
Record Dates: First submitted 2019-11-05; First posted 2019-11-13 (Actual); Last update posted 2021-11-08 (Actual); Status verified 2021-11

CONDITIONS: Urinary Disorders; Urinary Incontinence; Urinary Bladder Diseases
Keywords: Urodynamic; bladder; detrusor; urinary disorder
MeSH Terms: conditions — Urinary Incontinence; Urinary Bladder Diseases

STUDY DESIGN:
Intervention Model Description: NIRS module recording
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NIRS module (Experimental): Each patient has a NIRS module during a diagnosis urodynamic assessment provided for by the usual practice.
  Interventions: Device: NIRS recording

INTERVENTIONS:
Device: NIRS recording — Patient has a NIRS module during their urodynamic exam.

SUMMARY:
NIRS technology is therefore a technique that exploits the different absorption properties of oxygenated and deoxygenated hemoglobin to evaluate the degree of tissue oxygenation. This hemodynamic response is measured in a completely non-invasive and silent manner, by the simple emission of light passing through different layers of biological tissue.

In the literature, some studies concerning the use of the NIRS method for the study of urodynamics exist. They seem to show a correlation between the data of the urodynamic assessment and the data obtained with the NIRS method. Certain trends seem to be repeated with, for example, an increase in oxyhemoglobin at the beginning of the filling phase and the beginning of the urination phase.

The aim of the study is to analyze the NIRS signal and find correlation with urodynamic data.

DETAILED DESCRIPTION:
The main objective is to detect a urodynamic variation of the detrusor muscle during a contraction.

ELIGIBILITY:
Inclusion Criteria:

* Person whose urodynamic evaluation for diagnosis purposes is necessary
* Male or female ≥ 18 years
* Person affiliated with a social security scheme
* ECBU / BU negative

Exclusion Criteria:

* Minors
* Pregnant or parturient or lactating women
* Refusal of consent
* Contraindications usually provided for the realization of a Urodynamic exam
* Sensory disturbances making the participant insensitive to pain
* Motor or mental disorders that prevent the participant from expressing pain
* Behavioral problems that make the participant excessively agitated or aggressive
* Irritation and / or erythema, or open sore in the area covered by the NIRS
* Half-sitting position impossible
* Tattoo or stretch mark in the lower abdomen or pubic area
* External cutaneous or internal scar in the area covered by the NIRS
* Allergy to a component of the textile part of the device: polyamide, cotton, polyester, elastane, silver, other synthetic materials
* Simultaneous participation in another search

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — half of women and half of men
Enrollment: 40 (Actual)
Dates: Start 2020-07-07 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
optical measurement of hemoglobin concentrations | 9 months
  concentrations of oxygenated O2Hb, provided from a NIRS module
detrusor pressure measurement (Pdet) | 1 hour
  Pdet during filling and emptying of the urodynamic exam
optical measurement of hemoglobin concentrations | 9 months
  concentrations of deoxygenated HHb, provided from NIRS module
optical measurement of hemoglobin concentrations | 9 months
  concentrations of total tHB provided from NIRS module

SECONDARY OUTCOMES:
optical measurement of hemoglobin concentrations | 9 months
  concentrations of oxygenated O2Hb, provided from NIRS module
detrusor pressure measurement (Pdet) | 1 hour
  Pdet during filling and emptying of the urodynamic exam
optical measurement of hemoglobin concentrations | 1 hour
  concentrations of deoxygenated HHb, provided from NIRS module
clinical annotations of the doctor performed on the report of the urodynamic exam | 1 hour
  Normality of detrusor function (YES/NO), hyperactive detrusor function (YES/NO) , hypoactive detrusor function (YES/NO).
  Criteria assessed by the investigator by a response (yes/No)
optical measurement of hemoglobin concentrations | 9 months
  concentrations of total tHB provided from NIRS module

CONTACTS AND LOCATIONS:
Locations (1):
- Rangueil Hospital, Toulouse, France

IPD SHARING:
Plan to Share IPD: No